CLINICAL TRIAL: NCT04880135
Title: Effects of Supervised Versus Home Based Stretching and Strengthening Exercise Program on Neck Pain and Back Pain Among University Students Due to Quarantine During COVID-19: A Randomised Controlled Trial
Brief Title: Supervised Versus Home Based Exercises Neck and Low Back Pain Among Students Due to Quarantine During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00232
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal Pain; COVID-19; strengthening exercises; stretching exercises
MeSH Terms: conditions — Musculoskeletal Pain; COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised stretching and strengthening exercise (Experimental): Stretching and strengthening exercises will be performed under the supervision of Physical therapist for a period of one month
  Interventions: Other: Supervised stretching and strengthening exercise
- Home-based stretching and strengthening exercises (Experimental): Stretching and strengthening exercises will be performed at home by individuals having musculoskeletal pain due to quarantine for a period of one month.
  Interventions: Other: Home-based stretching and strengthening exercise

INTERVENTIONS:
Other: Supervised stretching and strengthening exercise — The structure of the supervised exercise sessions was a warm- up, followed by strengthening and finally stretching. Strengthening exercises will consist of a simple fitness plan of overhead press, push, pull and squat to stand which consist of 4 sets of 15 repetitions while stretching exercises protocol will be duration will be 4 sets of 10 repetitions. The total duration of the protocol will be of 50 to 60 minutes which consists of 10 minutes of warm up, strengthening for 20 to 25 minutes and stretching exercises for 15 to 20 minutes.
  Other Names: Rehabilitation following Supervised stretching and strengthening exercise
  Arms: Supervised stretching and strengthening exercise
Other: Home-based stretching and strengthening exercise — The structure of the home based exercise sessions was a warm- up, followed by strengthening and finally stretching. Strengthening exercises will consist of a simple fitness plan of overhead press, push, pull and squat to stand which consist of 4 sets of 15 repetitions while stretching exercises protocol will be duration will be 4 sets of 10 repetitions. The total duration of the protocol will be of 50 to 60 minutes which consists of 10 minutes of warm up, strengthening for 20 to 25 minutes and stretching exercises for 15 to 20 minutes.
  Other Names: Rehabilitation following Home-based stretching and strengthening exercise
  Arms: Home-based stretching and strengthening exercises

SUMMARY:
This study investigates whether or not the stretching and strengthening exercises are effective both at home and under supervision for people suffering from neck pain from using equipment for online courses due to quarantine during COVID-19.

DETAILED DESCRIPTION:
The aim of this study is to investigate which regime is best to follow a recommendation, be it under the supervision of the therapist or at home with stretching and strengthening exercises. There was no study that could explain the effect of stretching and strengthening exercises as a comparison between a supervised and a home treatment plan for neck pain in students during quarantine due to Covid-19.This study examines whether or not the recommendations given are effective both at home and under supervision.

ELIGIBILITY:
Inclusion Criteria

* Participants using gadget like computer, mobile or laptop for online education during quarantine
* Participants having musculoskeletal pain during COVID-19 quarantine
* Prolonged sitting and low physical activity during quarantine
* Prolonged exposure of screen more than 6 hours per day due online classes during the quarantine

Exclusion Criteria:

* Participants having musculoskeletal pain before the quarantine
* Participants doing any type of physical activity during quarantine
* Participants taking online classes or any online educational program before quarantine
* Participants with known congenital, inflammatory and infectious conditions of spine
* Participants following any ergonomic recommendations or any postural awareness during and after quarantine

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 month
  The visual analogue scale is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain ever with a frowning face image. 0 indicates no pain while 10 is worst pain.
International Physical Activity Questionnaire | 2 months
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available.
Neck Disability Index | 2 months
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life
Oswestry Low Back Pain Disability Questionnaire | 2 months
  Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. Questionnaire examines perceived level of disability in 10 everyday activities of daily living.
  The 6 statements are scored from 0 to 5 with the first statement scoring 0 through to the last at 5
Nordic Musculoskeletal Questionnaire | 2 months
  Nordic Musculoskeletal Questionnaire was used to provide the level of musculoskeletal pain from the previous 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No